CLINICAL TRIAL: NCT00384605
Title: A Phase III Randomized, Placebo-Controlled Clinical Trial to Study the Safety and Efficacy of Taranabant (MK0364) in Obese Patients and in Overweight Patients With Obesity-Related Co-Morbidities, Followed by a 1-Year Extension
Brief Title: An Investigational Drug Study to Assess Weight Loss in Obese and Overweight Patients (0364-037)(TERMINATED)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The overall profile does not support development for obesity
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0364-037; 2006_513
Record Dates: First submitted 2006-10-03; First posted 2006-10-06 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — N-(3-(4-chlorophenyl)-2-(3-cyanophenyl)-1-methylpropyl)-2-methyl-2-((5-(trifluoromethyl)pyridin-2-yl)oxy)propanamide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental): Arm 1: MK0364 2 mg capsule once daily
  Interventions: Drug: taranabant
- 2 (Experimental): Arm 2: MK0364 1 mg capsule once daily
  Interventions: Drug: taranabant
- 3 (Experimental): Arm 3: MK0364 0.5 mg capsule once daily.
  Interventions: Drug: taranabant
- 4 (Placebo Comparator): Arm 4: Pbo capsule once daily.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: taranabant — taranabant 0.5 mg capsule, 1 mg capsule, 2 mg capsule once daily. Treatment for 52 weeks.
  Arms: 1; 2; 3
Drug: placebo — Placebo capsule once daily. Treatment for 52 weeks.
  Arms: 4

SUMMARY:
A 1 year worldwide study in obese and overweight patients to assess the safety and effect on body weight of an investigational weight loss drug.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older, with Body Mass Index (BMI) between 30 kg/m2 and 43 kg/m2, inclusive (BMI between 27 kg/m2 and 43 kg/m2, inclusive, for those with obesity-related comorbidities). Obesity-related comorbidities associated with a BMI of 27 kg/m2 or higher include hypertension, dyslipidemia or sleep apnea
* Stable weight (+/-3 kg) for at least 3 months prior to study start

Exclusion Criteria:

* History of diabetes mellitis, major psychiatric disorder, significant cardiovascular disease, stroke, TIA, neurological disorder, non-febrile seizures
* Screening systolic blood pressure > 160 mm Hg or diastolic blood pressure > 100 mm Hg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2006-10; Primary Completion 2008-01 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Body weight after 52 weeks of treatment | 52 weeks

SECONDARY OUTCOMES:
Waist circumference, percent body fat, biochemical markers, blood pressure, and patient-reported outcomes after 52 weeks of treatment | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC